CLINICAL TRIAL: NCT05451446
Title: The Effect of Proprietary Water on Physiological and Perceptual Responses in Activities of Daily Living and a Heat Stressful Environment
Brief Title: The Effect of Proprietary Water on Physiological and Perceptual Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: HydraVes Technologies Inc. (Unknown)
Responsible Party: Principal Investigator, Susan Yeargin, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00112790
Record Dates: First submitted 2022-06-07; First posted 2022-07-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Hydration; Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Intervention Model Description: Between subjects, single-blind
Who Masked: Participant
Masking Description: Single-blind participants. They will not be told which group they are randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- proprietary water (Experimental): Participants in this group will consume a proprietary water blend for 5-free living days and then throughout their heat stress environment day.
  Interventions: Dietary Supplement: proprietary water
- carbohydrate-electrolyte drink (Active Comparator): Participants in this group will consume a commercial carbohydrate-electrolyte drink for 5-free living days and then throughout their heat stress environment day.
  Interventions: Other: Active comparator
- distilled water (Placebo Comparator): Participants in this group will consume distilled water for 5-free living days and then throughout their heat stress environment day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: proprietary water — They are randomized to consume a proprietary water product for five-free living days and to drink on the heat stress chamber day.
  Arms: proprietary water
Other: Active comparator — They are randomized to consume a carbohydrate drink for five-free living days and to drink on the heat stress chamber day.
  Arms: carbohydrate-electrolyte drink
Other: Placebo — They are randomized to consume water for five-free living days and to drink on the heat stress chamber day.
  Arms: distilled water

SUMMARY:
The purpose of this study is to determine if drinking proprietary water (PW) during a standardized daily plan as compared to distilled water (control) and carbohydrate-electrolyte (CE) drink can improve hydration status over time. Another purpose is to determine if PW, as compared to control and CE, can improve hydration status, perceptual responses, physiological responses, and cognition measures in a heat stressful environment. Healthy, physically active males and females aged 18 to 50y will be recruited for the study. Participants will be randomized into one of three groups: PW, CE, or Control. The participant will be given a daily standardized plan integrating their assigned fluid into daily hydration habits for five days. Participants will provide their first-morning urine sample, keep a daily food log, and answer questions about their perceptions of hydration. After the five days, they will participate in a treadmill exercise protocol within a warm environment (heat chamber). Multiple physiological, perceptual, and cognitive measures will be obtained while participants exercise and then recover.

DETAILED DESCRIPTION:
The study will investigate the effects of drinking proprietary water over a five-day free-living period and then during a heat stress environment compared to distilled water and a carbohydrate-electrolyte drink on markers of hydration, performance, and cognition. This will be a single-blind between-subjects study design. Participants will report to The University of South Carolina for two visits. At the first visit, potential participants will be explained the procedures and risks of the study and then sign an informed consent. Anthropometrics and demographic data will next be collected. Lastly, participants will be familiarized with specific measures and the testing protocol. Participants will take home study products to consume over 5-free living days in which they will need to keep a food and drink log and collect their first urine void of the day to drop off at the laboratory. After the free-living days, participants will return to the laboratory for their heat stress environment test. They will consume a standardized breakfast, complete questionnaires, then perform a 45-minute exercise protocol in the heat chamber. After the first 45-minutes, there will be a break to complete cognitive measures and return to the heat chamber for another 45-minute exercise protocol. Throughout the exercise protocols, participants will be responding to perceptual questions and blood draws. Following, they will rest for 60 minutes, during which they will answer more perceptual questionnaires and blood measures.

ELIGIBILITY:
Inclusion Criteria:

* regularly completing aerobic exercise (at least 3 times a week for >150 minutes/week) in order to complete the estimated 12K in the study protocol

Exclusion Criteria:

* current musculoskeletal injury restricting normal physical activity
* a "no" on the PAR-Q
* allergy to food dyes
* previous heat illness in the last year
* pregnancy
* any condition that could make exercising in warm conditions not safe (diabetes, cancer, etc.)
* certain medications (affecting blood pressure during exercise or hydration status)
* contraindications to the temperature pill

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Changes in plasma osmolality as a marker of hydration status. | On heat stress environment day. TP 2 (60 minutes).TP 5 (165 minutes). TP 7 (225 minutes).
  To determine if proprietary water has any effect on plasma osmolality compared to an active comparator and placebo.
Changes in core body temperature measured by ingestible telemetric pills or rectal thermometer. | On heat stress environment day. TP 1 (0 minute). TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes). Every 10-minutes during the exercise protocol.
  To determine if proprietary water has any effect on core body temperatures compared to an active comparator and placebo.
Changes in heart rate. | On heat stress environment day. TP 1 (0 minute). TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes). Every 10-minutes during the exercise protocol.
  To determine if proprietary water has any effect on heart rate compared to an active comparator and placebo.
Changes in urine specific gravity (USG) as a clinical marker of hydration status. | Every morning of the 5 free living days and TP 1(0 minute) on the heat stress day.
  To determine if proprietary water has any effect on USG compared to an active comparator and placebo.
Changes in plasma volume measured by hematocrit and hemoglobin | On heat stress environment day. TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes).
  To determine if proprietary water has any effect on plasma volume changes as compared to an active comparator and placebo.
Changes in sweat rate as measured by body mass changes. | On heat stress environment day. TP 1 (0 minute). TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes).
  To determine if proprietary water has any effect on sweat rate compared to an active comparator and placebo. This will be measured by body mass changes divided by the activity time.
Changes in thirst sensation | Every morning of the 5 free living days and on the heat stress day time points; TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes). 22:30 minute into 1st and 2nd 45 minute exercise
  To determine if proprietary water has any effect on thirst sensation assessed by a 9-point scale on Thirst Sensation, compared to an active comparator and placebo. The min score is 1 and the max score is 9, with higher scores associated with worse outcomes.
Changes in thermal sensation | Every morning of the 5 free living days and on the heat stress day time points; TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes). 22:30 minute into 1st and 2nd 45 minute exercise
  To determine if proprietary water has any effect on thirst sensation assessed by an 8-point scale on Thermal Sensation, compared to an active comparator and placebo. The min score is 0 and the max score is 8, with higher scores associated with worse outcomes.
Changes in slosh sensation | Every morning of the 5 free living days and on the heat stress day time points; TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes). 22:30 minute into 1st and 2nd 45 minute exercise
  To determine if proprietary water has any effect on thirst sensation assessed by a 9-point scale on Slosh Sensation, compared to an active comparator and placebo. The min score is 1 and the max score is 9, with higher scores associated with worse outcomes.
Changes in rating of perceived exertion | Every morning of the 5 free living days and on the heat stress day time points; TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes). 22:30 minute into 1st and 2nd 45 minute exercise
  To determine if proprietary water has any effect on thirst sensation assessed by Borgs RPE Scale, compared to an active comparator and placebo. The min score is 6 and the max score is 20, with higher scores associated with worse outcomes.
Changes in tension | Every morning of the 5 free living days and on the heat stress day time points; TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes).
  To determine if the proprietary water has an impact on tension-anxiety (POMS sub-score) compared to placebo and active comparator. Min 0, max 36, higher scores are associated with worse outcomes.
Changes in fatigue | Every morning of the 5 free living days and on the heat stress day time points; TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes).
  To determine if the proprietary water has an impact on fatigue (POMS sub-score) compared to placebo and active comparator. Min 0, max 28, higher scores are associated with worse outcomes.
Changes in anger | Every morning of the 5 free living days and on the heat stress day time points; TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes).
  To determine if the proprietary water has an impact on anger (POMS sub-score) compared to placebo and active comparator. Min 0, max 48, and higher scores are associated with worse outcomes.
Changes in depression | Every morning of the 5 free living days and on the heat stress day time points; TP 2 (60 minutes). TP 3 (105 minutes). TP 4 (125 minutes). TP 5 (165 minutes). TP 6 (195 minutes). TP 7 (225 minutes).
  To determine if the proprietary water has an impact on depression (POMS sub-score) compared to placebo and active comparator. Min 0, max 60, higher scores are associated with worse outcomes.
Changes in antidiuretic hormone (ADH) | On heat stress environment day. TP 2 (60 minutes).TP 5 (165 minutes). TP 7 (225 minutes).
  To determine if proprietary water has any effect on antidiuretic hormone (ADH) compared to an active comparator and placebo.
Changes in cortisol | On heat stress environment day. TP 2 (60 minutes).TP 5 (165 minutes). TP 7 (225 minutes).
  To determine if proprietary water has any effect on cortisol compared to an active comparator and placebo.
Changes in lactate | On heat stress environment day. TP 2 (60 minutes).TP 5 (165 minutes). TP 7 (225 minutes).
  To determine if proprietary water has any effect on lactate compared to an active comparator and placebo.

SECONDARY OUTCOMES:
Changes in object hit and avoid | Baseline day 0 and on heat stress environment day 5 timepoints: TP 1 (0 minute). TP 3 (105 minutes). TP 5(165 minutes).
  To determine if proprietary water has any effect on cognitive task of "object hit and avoid" compared to an active comparator and placebo.
Changes in trail making task | Baseline day 0 and on heat stress environment day 5 timepoints: TP 1 (0 minute). TP 3 (105 minutes). TP 5(165 minutes).
  To determine if proprietary water has any effect on cognitive task of "trail making task" compared to an active comparator and placebo.
Changes in N-Back task | Baseline day 0 and on heat stress environment day 5 timepoints: TP 1 (0 minute). TP 3 (105 minutes). TP 5(165 minutes).
  To determine if proprietary water has any effect on cognitive task of "N-Back Task" compared to an active comparator and placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina Sport Science Lab, Columbia, South Carolina, United States